CLINICAL TRIAL: NCT01599104
Title: A Multi-center, Randomized, Double-blind, Active-controlled, 8-week Study to Evaluate the Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Japanese Patients With Essential Hypertension
Brief Title: Efficacy and Safety of LCZ696 in Comparison to Olmesartan in Japanese Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696A1306
Record Dates: First submitted 2012-05-13; First posted 2012-05-15 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; LCZ696
MeSH Terms: conditions — Essential Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; olmesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LCZ696 200 mg (Experimental): LCZ696 200 mg tablet and placebo to both LCZ696 (1 tablet) and Olmesartan (1 capsule) tablet once daily for 8 weeks
  Interventions: Drug: LCZ696; Drug: Placebo
- LCZ696 400 mg (Experimental): LCZ696 200 mg tablet and a placebo to both LCZ696 (1 tablet) and Olmesartan (1 capsule) once daily for one week; then up-titrated to LCZ696 400 mg and placebo to Olmesartan (1 capsule) once daily for the remaining 7 weeks
  Interventions: Drug: LCZ696; Drug: Placebo
- Olmesartan 20 mg (Active Comparator): Olmesartan 20 mg capsule and placebo to LCZ696 (2 tablets) once daily for 8 weeks
  Interventions: Drug: Olmesartan; Drug: Placebo

INTERVENTIONS:
Drug: LCZ696 — 200 mg (one tablet) or 400 mg (2 tablets of 200mg) once daily
  Arms: LCZ696 200 mg; LCZ696 400 mg
Drug: Olmesartan — Olmesartan 20 mg capsule one daily
  Arms: Olmesartan 20 mg
Drug: Placebo — Placebo to LCZ696 or Olmesartan

SUMMARY:
This study assessed the efficacy of LCZ696 in Japanese patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-to-moderate hypertension, untreated or currently taking antihypertensive therapy.
* Treated patients (using antihypertensive treatments within 4 weeks prior to Visit 1) must have an msSBP ≥ 150 mmHg and < 180 mmHg at the randomization visit (Visit 201) and msSBP ≥140 mmHg < 180 mmHg at the visit immediately proceeding Visit 201 (Visit 102 or 103).
* Untreated patients (newly diagnosed with essential hypertension or having a history of hypertension but have not been taking any antihypertensive drugs for at least 4 weeks prior to Visit 1) must have an msSBP ≥ 150 mmHg and < 180 mmHg at both Visit 1 and Visit 201.
* Patients must have an absolute difference of ≤15 mmHg in msSBP between Visit 201 and the immediately preceding visit;

Exclusion Criteria:

* Severe hypertension (msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg).
* History of angioedema, drug-related or otherwise, as reported by the patient.
* History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension.
* Patients who previously entered a LCZ696 study and had been randomized or enrolled into the active drug treatment epoch.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- Japan (42):
  - Novartis Investigative Site, Kamogawa, Chiba
  - Novartis Investigative Site, Chikushi-gun, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Kyōtanabe, Kyoto
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Ibadraki, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Fujimino, Saitama
  - Novartis Investigative Site, Hiki-Gun, Saitama
  - Novartis Investigative Site, Koshigaya, Saitama
  - Novartis Investigative Site, Niiza, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Sakado, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Kunitachi, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shibuya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Tachikawa, Tokyo
  - Novartis Investigative Site, Taitō City, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo

REFERENCES:
- [Derived] Kario K, Rakugi H, Yarimizu D, Morita Y, Eguchi S, Iekushi K. Twenty-Four-Hour Blood Pressure-Lowering Efficacy of Sacubitril/Valsartan Versus Olmesartan in Japanese Patients With Essential Hypertension Based on Nocturnal Blood Pressure Dipping Status: A Post Hoc Analysis of Data From a Randomized, Double-Blind Multicenter Study. J Am Heart Assoc. 2023 Apr 18;12(8):e027612. doi: 10.1161/JAHA.122.027612. Epub 2023 Apr 7. PMID 37026551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of 3 epochs: 1)screening, 2) single blind run-in and 3) double blind treatment. During the run-in epoch, eligible participants received placebo to both treatments for 2 to 4 weeks. After the run-in epoch, a total of 1161 eligible participants continued into the double blind treatment epoch for 8 weeks.
Groups:
- LCZ696 200 mg: LCZ696 200 mg tablet and a placebo tablet once daily for eight weeks
- LCZ696 400 mg: LCZ696 200 mg tablet and a placebo tablet once daily for one week, then up-titrated to 400 mg once daily for the remaining 7 weeks
- Olmesartan 20 mg: Olmesartan 20 mg tablet and a placebo tablet once daily for 8 weeks
Period: Overall Study
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Started | 387 | 385 | 389
Completed | 371 | 371 | 363
Not Completed | 16 | 14 | 26
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Technical Problems | 1 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 2
Not completed — Non-compliance with study treatment | 0 | 1 | 0
Not completed — Lack of Efficacy | 4 | 4 | 10
Not completed — Adverse Event | 7 | 6 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg | Total
Number analyzed (Participants) | 387 | 385 | 389 | 1161
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (10.87) | 58.7 (10.50) | 59.6 (10.50) | 58.7 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 117 | 103 | 343
  Male | 264 | 268 | 286 | 818

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: Sitting BP measurements were performed at screening through the end of study at every visit. Four separate sitting BP were obtained with a full two-minute interval between measurements. The 4 measurements were summed and averaged, and then the baseline BP value was subtracted from the average value to get the change from baseline.
Time Frame: Baseline, 8 weeks
Population: Full Analysis Set (FAS): The full analysis set included all randomized participants who received study medication and had both baseline and post-baseline BP assessments.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
mmHg | -18.21 (0.702) | -20.18 (0.704) | -13.20 (0.700)

2. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory SBP (maSBP) at Week 8
Description: Ambulatory blood pressure monitoring (ABPM) over a 24-hour period was conducted at two time-points during the study in a subset of participants.
Time Frame: Baseline, 8 weeks
Population: The full analysis set included all randomized participants who received study medication, and had both baseline and post-baseline ABPM measurements. This outcome measure was analyzed in a subset of participants within each treatment group where n = 216 for the LCZ 200 mg group, n = 216 for the LCZ 400 mg group and n = 200 for the Olmesartan group.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 216 | 216 | 200
mmHg | -13.44 (0.445) | -14.99 (0.445) | -8.78 (0.462)

3. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Sitting BP measurement was performed at screening through the end of study at every visit. Four separate sitting BP were obtained with a full two-minute interval between measurement. The 4 measurements were summed and averaged, and then the baseline BP value was subtracted from the average value to get the change from baseline.
Time Frame: Baseline, 8 weeks
Population: The full analysis set included all randomized participants who received study medication, and had both baseline and post-baseline BP measurements.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
mmHg | -7.76 (0.404) | -8.79 (0.406) | -5.91 (0.404)

4. Secondary Outcome: Percentage of Participants Achieving a Successful Response in Overall Blood Pressure Control at Week 8
Description: A successful response in overall BP control rate was defined as msSBP < 140 mmHg and msDBP <90 mmHg.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
Percentage of participants | 43.9 | 46.5 | 32.9

5. Secondary Outcome: Percentage of Participants Achieving a Successful msSBP Response
Description: Successful msSBP response was defined as < 140 mmHg or ≥ 20 mmHg reduction from baseline.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
Percentage of participants | 57.9 | 63.1 | 42.9

6. Secondary Outcome: Percentage of Participants Achieving a Successful msDBP Response
Description: Successfull msDBP response was defined as <90 mmHg or ≥10 mmHg reduction from baseline.
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
Percentage of participants | 69.5 | 70.1 | 60.7

7. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory DBP (maDBP) at Week 8
Description: ABPM over a 24-hour period was conducted at two time-points during the study in a subset of participants.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 216 | 216 | 200
mmHg | -7.65 (0.295) | -8.44 (0.295) | -5.56 (0.307)

8. Secondary Outcome: Change From Baseline in maSBP and maDBP for Daytime/Nighttime
Description: ABPM over a 24-hour period was conducted at two time-points during the study in a subset of participants.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 216 | 216 | 200
mmHg
  maSBP daytime | -12.60 (0.747) | -14.44 (0.747) | -7.87 (0.776)
  maSBP nighttime | -15.13 (0.747) | -16.09 (0.747) | -10.65 (0.776)
  maDBP daytime | -7.01 (0.506) | -8.00 (0.506) | -4.95 (0.526)
  maDBP nighttime | -8.82 (0.506) | -9.42 (0.506) | -6.79 (0.526)

9. Secondary Outcome: Change From Baseline in Office Pulse Pressure
Description: Office pulse pressure was calculated as msSBP minus msDBP. Sitting blood pressure (BP) measurement was performed at screening through the end of study at every visit. Four separate sitting BP were obtained with a full two-minute interval between measurement. The 4 measurements were summed and then averaged to calculate the mean BP value. The baseline PP value was subtracted from the week 8 PP value to determine the change from baseline in PP.
Time Frame: Baseline, 8 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
mmHg | -10.49 (0.471) | -11.30 (0.472) | -7.34 (0.470)

10. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Pulse Pressure
Description: Ambulatory pulse pressure was calculated as hourly ambulatory SBP minus hourly ambulatory DBP in a subset of participants.
Time Frame: Baseline, 8 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 216 | 216 | 200
mmHg | -5.79 (0.208) | -6.57 (0.207) | -3.20 (0.216)

11. Secondary Outcome: Number of Patients With Adverse Events, Serious Adverse Events and Death
Description: Participants were monitored for adverse events, serious adverse events and deaths throughout the study.
Time Frame: 8 weeks
Population: Safety Set. The safety set included aqll participants who had received study medication.
Measure: Number; unit: Participants
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Number analyzed (Participants) | 387 | 385 | 389
Participants
  Adverse Events (serious and non-serious) | 135 | 136 | 152
  Seroius Adverse Events | 1 | 1 | 7
  Deaths | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | LCZ696 200 mg | LCZ696 400 mg | Olmesartan 20 mg
Serious Adverse Events (participants affected / at risk) | 1/387 | 1/385 | 7/389
Other Adverse Events (participants affected / at risk) | 48/387 | 47/385 | 46/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=387) | LCZ696 400 mg (N=385) | Olmesartan 20 mg (N=389)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
CATARACT (Eye disorders) | 0 | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 1
HEPATOBILIARY DISEASE (Hepatobiliary disorders) | 0 | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 1
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 200 mg (N=387) | LCZ696 400 mg (N=385) | Olmesartan 20 mg (N=389)
NASOPHARYNGITIS (Infections and infestations) | 48 | 47 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.